CLINICAL TRIAL: NCT05881421
Title: Prospective Multi-Center, Post-Market, Observational Study (OS) of the Shockwave Medical, Inc. Intravascular Lithotripsy System in Peripheral Arteries
Brief Title: DISRUPT PAD III Observational Study
Acronym: PAD III OS
Status: Completed | Type: Observational
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 60892 OS
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Intravascular Lithotripsy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Disrupt PAD III study was designed as a randomized controlled trial (RCT) with an additional observational registry component. The registry, referred to as the Disrupt PAD III Observational Study (PAD III OS), was a global, prospective, multi-center, single-arm registry of the Shockwave Peripheral Intravascular Lithotripsy (IVL) System. The objective of this study was to assess the real-world acute performance of IVL in the treatment of calcified, stenotic, peripheral arteries that may not qualify for inclusion in the RCT. The study was designed to enroll a maximum of 1500 subjects from up to 60 global sites with a minimum of 200 subjects treated with the S4 IVL catheter, a line extension designed to treat smaller diameter peripheral vessels, including calcified below-the-knee (BTK) lesions.

Subjects were required to have target lesions in the iliac, femoral, ilio-femoral, popliteal, or infra-popliteal arteries with at least moderate calcification as determined by the investigator, defined as calcification within the lesion on both sides of the vessel assessed by angiography. Adjunctive therapies such as atherectomy, specialty balloons, and stents were allowed. Subjects were followed through discharge.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to meet ALL of the following inclusion criteria in order to be included in this clinical study:

1. Subjects intended to be treated with Shockwave Medical Lithoplasty for de-novo or restenotic lesions of the femoral, ilio-femoral, popliteal, and infra-popliteal arteries.
2. Subjects presenting with claudication or CLI by Rutherford Clinical Category 2, 3, 4, 5, or 6 of the target limb.
3. Age of subject is > 18.
4. Subject of subject's legal representative have been informed of the nature of the study, agrees to participate and has signed the approved consent form.
5. Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

Exclusion Criteria:

Subjects that met ANY of the following exclusion criteria were not included in this clinical study:

1. Subjects with any medical condition that would make him/her an inappropriate candidate for treatment with Shockwave Lithoplasty as per Instructions for Use (IFU) or investigator's opinion.
2. Subject already enrolled in other investigational (interventional) studies that would interfere with study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the study sites with known PAD requiring an interventional procedure were evaluated for eligibility and participation in the study. If a patient met the baseline pre-procedure screening of inclusion and none of the exclusion criteria for the protocol version current at time of screening, and was willing to participate in the study, written consent was obtained. No study-specific requirements were performed prior to obtaining informed consent.
Sampling Method: Probability Sample
Enrollment: 1373 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Procedural Success - Primary Effectiveness Endpoint | Peri-procedural, approximately 2 hours
  Defined as final residual stenosis ≤30% without flow-limiting dissection (≥ grade D) by angiographic core lab. In the primary analysis, Procedural Success was assessed on a per-subject basis; for subjects with multiple IVL-treated lesions, Procedural Success was achieved if all lesions met criteria.

SECONDARY OUTCOMES:
Procedural Success - Secondary Effectiveness Endpoint | Peri-procedural, approximately 2 hours
  As secondary analyses, Procedural Success was also assessed on a per-lesion basis, as well as using a <50% residual stenosis threshold.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (26):
  - Stanford Hospital, Palo Alto, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth Northern Colorado, Loveland, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Tallahassee Research Institute Inc., Tallahassee, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Steward St. Elizabeth's Medical Center, Brighton, Massachusetts
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Cardiovascular Consultants, Kansas City, Missouri
  - Mount Sinai West, New York, New York
  - Columbia University Medical Center, New York, New York
  - NC Heart & Vascular Research, LLC, Raleigh, North Carolina
  - Ohio Health Research Institute, Columbus, Ohio
  - St. John Clinic, Bartlesville, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pinnacle Health Cardiovascular Institute, Harrisburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Baptist Medical Center, Memphis, Tennessee
  - St. David's Heart and Vascular (Austin Heart), Austin, Texas
  - Baylor Clinic McNair Campus, Houston, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
- Germany (3):
  - Evangelisches Krankenhaus Mulheim an der Ruhr, Mülheim
  - St. Franziskus Hospital, Münster
  - RoMed Klinikum Rosenheim, Rosenheim
- Auckland City Hospital, Auckland, New Zealand